CLINICAL TRIAL: NCT00037115
Title: An Open Label Pilot Study of Induction Therapy With a Single High Dose Bolus of Intravenous Methotrexate With Leucovorin Rescue, Prior to Initiation of AVONEX® Treatment, in Patients Presenting With a First Acute Demyelinating Event: Comparison With CHAMPS Results.
Brief Title: Induction Therapy With a Single High Dose Bolus of Intravenous Methotrexate With Leucovorin Rescue, Prior to Initiation of AVONEX® Treatment, in Patients Presenting With a First Acute Demyelinating Event.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: MidAmerica Neuroscience Research Foundation at Rowe Neurology Institute (Other)
Collaborators: Consultants in Neurology (Industry)
Responsible Party: Principal Investigator, Vernon D. Rowe III, MD, Vernon D. Rowe III, MD, MidAmerica Neuroscience Research Foundation at Rowe Neurology Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MANI-MTX02-001
Record Dates: First submitted 2002-05-15; First posted 2002-05-17 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Demyelinating Disorders; Multiple Sclerosis; Optic Neuritis; Myelitis; Neuritis
Keywords: Demyelinating; Multiple Sclerosis; Myelitis; Neuritis; Optic Neuritis; AVONEX; methotrexate; methylprednisolone; interferon beta 1a; demyelination; central nervous system; brain; nerve; lesions; enhancement; enhancing
MeSH Terms: conditions — Demyelinating Diseases; Multiple Sclerosis; Optic Neuritis; Myelitis; Neuritis | interventions — Interferon beta-1a; Methotrexate; Methylprednisolone

INTERVENTIONS:
Drug: interferon beta 1a
Drug: methotrexate
Drug: methylprednisolone

SUMMARY:
The participant will receive weekly intramuscular treatment with AVONEX® (interferon beta 1-a) and a one-time high dose intravenous methotrexate with Leucovorin rescue, along with the standard solumedrol treatment before beginning AVONEX® treatment.

DETAILED DESCRIPTION:
The participant will receive weekly intramuscular treatment with AVONEX® (interferon beta 1-a) and a one-time high dose intravenous methotrexate with Leucovorin rescue, along with the standard solumedrol treatment before beginning AVONEX® treatment.

At study entrance, baseline lab work (complete blood count, platelet count, routine electrolytes, blood urea nitrogen, creatinine, liver function tests, 24 hour urine collection for creatinine clearance, urine pregnancy test, urinalysis and urine culture and sensitivity if needed), and an electrocardiogram (measurement of heart activity) will be done. A complete medical history, neurological and opthamological examination will be performed, including measurements of vital signs (heart rate and blood pressure), as well as magnetic resonance imaging (MRI), EDSS, and Visual Evoked Response test (VER's) to document status of disease. A Multiple Sclerosis Functional Composite Score (MSFC) consists of the Timed 25 Foot Walk, Nine Hole Peg Test (9HPT), and Paced Auditory Serial Addition Test 3 (PASAT3) will be performed at screen as well. At months 6, 12, 18, 24, 30 and 36 the tests and evaluations will include MRI, MSFC, VER's and blood tests of immune cells. Other safety evaluations (previously mentioned blood and urine tests) will be conducted according to the date of treatment. These tests include a laboratory test (methotrexate level) two days following treatment, as well as routine lab tests 2 weeks following the methotrexate treatment. This treatment would be under the supervision of Dr. Rowe.

The patients will continue their AVONEX® intramuscular injections of 30 micrograms (administered by patient or caregiver) on a weekly basis. The methylprednisolone treatment and methotrexate infusion will be performed in our outpatient infusion center. The patient will be required to complete a patient diary during the course of the trial, participate in and keep all scheduled appointments, and to inform the research staff and physician of any change in concomitant medications or adverse events that they may experience.

ELIGIBILITY:
To be eligible for entry into this study, candidates must meet the following eligibility criteria at the time of enrollment, which are the same as in the CHAMPS study [1]:

* Between the ages of 18 and 50 years, inclusive.
* As in the CHAMPS study [1] patients must have had a first isolated, well-defined neurologic event consistent with demyelination and involving the optic nerve (unilateral optic neuritis), spinal cord (incomplete transverse myelitis), or brain stem or cerebellum (brain stem or cerebella syndrome). They must also have two or more clinically silent lesions of the brain that were at least 3 mm in diameter on MRI scans and were characteristic of MS (at least one lesion must be periventricular or ovoid).
* The onset of the visual or neurological symptoms must have occurred no more than twelve days before the MTX treatment, so that the methylprednisolone treatment is begun no more than fourteen days after the onset of symptoms, as in CHAMPS.
* Patients must give written informed consent prior to any testing under this protocol, including screening tests and evaluations that are not considered part of the subject's routine care.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2002-05 (Actual); Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MidAmerica Neuroscience Institute, Kansas City, Missouri, United States